CLINICAL TRIAL: NCT05620485
Title: Timing of Operation in Children With a Prenatal Diagnosis of Choledochal Cyst：A Single-center Prospective Study
Brief Title: Timing of Operation in Children With a Prenatal Diagnosis of Choledochal Cyst
Acronym: CDCPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Xisi Guan, Clinical attending doctor, Guangzhou Women and Children's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 521123
Record Dates: First submitted 2022-10-02; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Choledochal Cyst
MeSH Terms: conditions — Choledochal Cyst

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prenatally diagnosed CDC (Experimental): All patients received laparoscopic-assisted CDC excision and hepaticojejunostomy.
  Interventions: Procedure: laparoscopic-assisted CDC excision and hepaticojejunostomy

INTERVENTIONS:
Procedure: laparoscopic-assisted CDC excision and hepaticojejunostomy — After birth, the liver and gallbladder ultrasound were regularly rechecked. If the maximum diameter of the cyst was greater than 5 cm, surgery was performed.

SUMMARY:
In this prospective study, we tried to select the operation time according to the cyst size and evaluate the treatment effect.

DETAILED DESCRIPTION:
A choledochal cyst (CDC) is a congenital anomaly of the biliary system, which is more common in the Asian population. If a CDC is not diagnosed and treated promptly, it often leads to a series of serious complications, including cholangitis, cyst rupture, cholestatic cirrhosis, and even cholangiocarcinoma. Infants with a postnatal diagnosis of CDC often present with symptoms, and to avoid the occurrence of serious complications, operative correction should be performed as soon as possible when their clinical conditions allow. However, in the current era with the improvement of prenatal screening technology, an increasing number of choledochal cysts are diagnosed prenatally in the fetus. In developed countries, as many as 15% of choledochal cysts are found before birth. Some of these children receive intervention when they are asymptomatic at an early stage, while some have progressed to CDC-related symptoms before operative correction. The timing of operation for children with a prenatal diagnosis of CDC remains controversial. The investigators previous study showed that it is more advantageous to receive surgical treatment in the asymptomatic period for patients with prenatally diagnosed CDC. In addition, the age at operation (months) appears to be unrelated to intraoperative and postoperative complications, which is distinct from previous studies. More interestingly, the investigators found that a specific cyst size (length > 5.2 cm and width > 4.1 cm) suggested that clinical symptoms might appear and that the surgery should be performed as soon as clinically safe to proceed. Therefore, in this study, the investigators tried to select the operation time according to the cyst size and evaluate the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with a prenatal and postnatal diagnosis with CDC
2. Prenatal and postnatal hepatobiliary ultrasound data were complete
3. Age of visit < 3 months

Exclusion Criteria:

Unable to tolerate surgery after birth

Ages: 0 Months to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
preoperative complications | pre-intervention
  number of participants progressed to CDC-related symptoms before operative intervention
preoperative complications | pre-intervention
  number of participants with cyst rupture before operative intervention
preoperative complications | 1 week before surgery
  aspartate aminotransferase (U/L)
preoperative complications | 1 week before surgery
  alanine aminotransferase (U/L)
preoperative complications | 1 week before surgery
  γ-glutamyl transpeptidase (U/L)
preoperative complications | 1 week before surgery
  Serum Bilirubin (μmol/L）
short-term complications | 1 weak after surgery
  number of participants with post-operative anastomotic leak
short-term complications | 1 weak after surgery
  number of participants with postoperative hemorrhage
short-term complications | 1 weak after surgery
  aspartate aminotransferase (U/L)
short-term complications | 1 weak after surgery
  alanine aminotransferase (U/L)
short-term complications | 1 weak after surgery
  γ-glutamyl transpeptidase (U/L)
short-term complications | 1 weak after surgery
  Serum Bilirubin (μmol/L）
short-term complications | 3 months after surgery
  aspartate aminotransferase (U/L)
short-term complications | 3 months after surgery
  alanine aminotransferase (U/L)
short-term complications | 3 months after surgery
  γ-glutamyl transpeptidase (U/L)
short-term complications | 3 months after surgery
  Serum Bilirubin (μmol/L）
short-term complications | 6 months after surgery
  aspartate aminotransferase (U/L)
short-term complications | 6 months after surgery
  alanine aminotransferase (U/L)
short-term complications | 6 months after surgery
  γ-glutamyl transpeptidase (U/L)
short-term complications | 6 months after surgery
  Serum Bilirubin (μmol/L）
short-term complications | 1 month after surgery
  number of participants with postoperative wound infection
Long-term complications | 3 years after surgery
  number of participants with anastomotic stricture

SECONDARY OUTCOMES:
length of stay | 1 month after surgery
  length of hospital stay
duration of ventilator support | 1 month after surgery
  duration of ventilator support
length of nutritional support in hospital | 1 month after surgery
  length of nutritional support in hospital

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-10-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT05620485/Prot_000.pdf